CLINICAL TRIAL: NCT01115283
Title: Improving Spatial and Temporal Vision in Adult and Juvenile Amblyopia
Brief Title: An Active Approach to Treat Amblyopia: Perceptual Learning and Video Games
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R01EY001728 (NIH); R01EY001728 (NIH)
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Amblyopia
Keywords: amblyopia treatment; neural plasticity; perceptual learning; vision therapy; spatial vision; video games; occlusion therapy
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perceptual learning (Experimental): Patients will be asked to practice a range of visual discrimination tasks for a period of time (each therapy session:1-2 hrs, 4-5 sessions/wk for ~1-6 months).
  Interventions: Behavioral: Perceptual learning
- Occlusion therapy (Experimental): The fellow sound will be covered with a standard eye patch for a period of time (1-2 hrs/day, 4-5 days/wk for ~1-3 months). The idea is to push the brain to use the weaker amblyopic eye.
  Interventions: Behavioral: Occlusion therapy
- Video game (Experimental): Patients will be asked to play videogames for a period of time (each therapy session:1-2 hrs, 4-5 sessions/wk for ~1-6 months).
  Interventions: Behavioral: Video Games

INTERVENTIONS:
Behavioral: Perceptual learning — Research participants will be asked to practice a visual discrimination task (e.g. position acuity, contrast sensitivity, stereoacuity etc) in our laboratory for a period of time (2 hrs/day, 5 days/week).
  Other Names: vision therapy; vision training
  Arms: Perceptual learning
Behavioral: Video Games — Research participants will be asked to play "off-the-shelf" video games in our laboratory for a period of time (2 hrs/day, 5 days/week).
  Other Names: vision therapy; vision training
  Arms: Video game
Behavioral: Occlusion therapy — Research participants will be required to cover the good eye during the day in order to push the brain to use the amblyopic eye (2 hrs/day, 5 days/week for 2-4 weeks).
  Other Names: vision training,; vision therapy
  Arms: Occlusion therapy

SUMMARY:
Amblyopia, a developmental abnormality that impairs spatial vision, is a major cause of vision loss, resulting in reduced visual acuity and reduced sensitivity to contrast. This study uses psychophysical measures to study neural plasticity in both adults and children with amblyopia.

DETAILED DESCRIPTION:
Amblyopia, a developmental abnormality that impairs spatial vision, is a major cause of vision loss, resulting in reduced visual acuity and reduced sensitivity to contrast. Our previous findings (see CITATIONS) show that the adult amblyopic brain is still plastic and malleable, suggesting that active approach is potential useful in treating amblyopia. The goal of this project is to assess the limits and mechanisms of neural plasticity in both normal and amblyopic spatial vision. This study uses psychophysical measures to study neural plasticity in both adults and children with amblyopia. Research participants will be asked to practice a visual discrimination task (perceptual learning) or to play video games with the amblyopic eye for a period of time. A range of visual functions will be monitored during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* adults and children (>5 years old) with normal vision or amblyopia
* amblyopia: interocular VA difference of at least 0.1 logMAR

Exclusion Criteria:

* any ocular pathological conditions, nystagmus

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Amblyopic vision | 9 months
  Improvement in amblyopic vision : visual acuity and stereoacuity

SECONDARY OUTCOMES:
Spatial vision | 9 months
  Improvement in spatial vision (eg. contrast sensitivity, positional acuity and spatial attention)
Temporal vision | 9 months
  Improvement in temporal processing and temporal vision

CONTACTS AND LOCATIONS:
Overall Officials: Roger W Li, OD, PhD, Principal Investigator — School of Optometry, Univeristy of california-Berkeley; Dennis M Levi, OD, PhD, Principal Investigator — School of Optometry, Univerisity of California-Berkeley
Locations (1):
- Minor Hall 486, School of Optometry, University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Background] Levi DM, Li RW. Improving the performance of the amblyopic visual system. Philos Trans R Soc Lond B Biol Sci. 2009 Feb 12;364(1515):399-407. doi: 10.1098/rstb.2008.0203. PMID 19008199
- [Background] Levi DM, Li RW. Perceptual learning as a potential treatment for amblyopia: a mini-review. Vision Res. 2009 Oct;49(21):2535-49. doi: 10.1016/j.visres.2009.02.010. Epub 2009 Feb 27. PMID 19250947
- [Background] Bavelier D, Levi DM, Li RW, Dan Y, Hensch TK. Removing brakes on adult brain plasticity: from molecular to behavioral interventions. J Neurosci. 2010 Nov 10;30(45):14964-71. doi: 10.1523/JNEUROSCI.4812-10.2010. PMID 21068299
- [Background] Chung ST, Kumar G, Li RW, Levi DM. Characteristics of fixational eye movements in amblyopia: Limitations on fixation stability and acuity? Vision Res. 2015 Sep;114:87-99. doi: 10.1016/j.visres.2015.01.016. Epub 2015 Feb 7. PMID 25668775
- [Background] Li RW, So K, Wu TH, Craven AP, Tran TT, Gustafson KM, Levi DM. Monocular blur alters the tuning characteristics of stereopsis for spatial frequency and size. R Soc Open Sci. 2016 Sep 21;3(9):160273. doi: 10.1098/rsos.160273. eCollection 2016 Sep. PMID 27703690
- [Result] Li RW, Klein SA, Levi DM. Prolonged perceptual learning of positional acuity in adult amblyopia: perceptual template retuning dynamics. J Neurosci. 2008 Dec 24;28(52):14223-9. doi: 10.1523/JNEUROSCI.4271-08.2008. PMID 19109504
- [Result] Li RW, Provost A, Levi DM. Extended perceptual learning results in substantial recovery of positional acuity and visual acuity in juvenile amblyopia. Invest Ophthalmol Vis Sci. 2007 Nov;48(11):5046-51. doi: 10.1167/iovs.07-0324. PMID 17962456
- [Result] Li RW, Young KG, Hoenig P, Levi DM. Perceptual learning improves visual performance in juvenile amblyopia. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3161-8. doi: 10.1167/iovs.05-0286. PMID 16123415
- [Result] Li RW, Levi DM. Characterizing the mechanisms of improvement for position discrimination in adult amblyopia. J Vis. 2004 Jun 1;4(6):476-87. doi: 10.1167/4.6.7. PMID 15330715
- [Result] Chung ST, Li RW, Levi DM. Identification of contrast-defined letters benefits from perceptual learning in adults with amblyopia. Vision Res. 2006 Oct;46(22):3853-61. doi: 10.1016/j.visres.2006.06.014. Epub 2006 Aug 22. PMID 16930666
- [Result] Chung ST, Li RW, Levi DM. Learning to identify near-threshold luminance-defined and contrast-defined letters in observers with amblyopia. Vision Res. 2008 Dec;48(27):2739-50. doi: 10.1016/j.visres.2008.09.009. Epub 2008 Oct 18. PMID 18824189
- [Result] Li RW, Ngo CV, Levi DM. Relieving the attentional blink in the amblyopic brain with video games. Sci Rep. 2015 Feb 26;5:8483. doi: 10.1038/srep08483. PMID 25715870
- [Result] Chung ST, Li RW, Levi DM. Learning to identify near-acuity letters, either with or without flankers, results in improved letter size and spacing limits in adults with amblyopia. PLoS One. 2012;7(4):e35829. doi: 10.1371/journal.pone.0035829. Epub 2012 Apr 30. PMID 22558234
- [Result] Li RW, Ngo C, Nguyen J, Levi DM. Video-game play induces plasticity in the visual system of adults with amblyopia. PLoS Biol. 2011 Aug;9(8):e1001135. doi: 10.1371/journal.pbio.1001135. Epub 2011 Aug 30. PMID 21912514
- [Result] Li RW, Tran TT, Craven AP, Leung TW, Chat SW, Levi DM. Sharpening coarse-to-fine stereo vision by perceptual learning: asymmetric transfer across the spatial frequency spectrum. R Soc Open Sci. 2016 Jan 20;3(1):150523. doi: 10.1098/rsos.150523. eCollection 2016 Jan. PMID 26909178
- [Result] Chung STL, Li RW, Silver MA, Levi DM. Donepezil Does Not Enhance Perceptual Learning in Adults with Amblyopia: A Pilot Study. Front Neurosci. 2017 Aug 7;11:448. doi: 10.3389/fnins.2017.00448. eCollection 2017. PMID 28824369
- [Result] Li RW, Tran KD, Bui JK, Antonucci MM, Ngo CV, Levi DM. Improving Adult Amblyopic Vision with Stereoscopic 3-Dimensional Video Games. Ophthalmology. 2018 Oct;125(10):1660-1662. doi: 10.1016/j.ophtha.2018.04.025. Epub 2018 May 18. No abstract available. PMID 29779684
- [Result] Levi DM, Li RW, Silver MA, Chung STL. Sequential perceptual learning of letter identification and "uncrowding" in normal peripheral vision: Effects of task, training order, and cholinergic enhancement. J Vis. 2020 Apr 9;20(4):24. doi: 10.1167/jov.20.4.24. PMID 32347910
- [Derived] Godinez A, Martin-Gonzalez S, Ibarrondo O, Levi DM. Scaffolding depth cues and perceptual learning in VR to train stereovision: a proof of concept pilot study. Sci Rep. 2021 May 12;11(1):10129. doi: 10.1038/s41598-021-89064-z. PMID 33980895